CLINICAL TRIAL: NCT05307224
Title: The Effect of Mandala Painting on Anxiety in Coronary Heart Patients: A Randomized Controlled Trial
Brief Title: The Effect of Mandala Painting on Anxiety in Coronary Heart Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Gülşah Çamcı, Assistant Prof, Marmara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MU-SBF-IHH-GC-02
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease; Anxiety
Keywords: Coronary Artery Disease; Anxiety; mandala
MeSH Terms: conditions — Coronary Artery Disease; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: control group (usual care) and experimental group (mandala painting)
Who Masked: Participant
Masking Description: It was planned to use block randomization for the random assignment of patients to the experimental and control groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In the experimental group, patients will receive both routine care and mandala painting. Experimental group will paint mandala for 30 minutes/day in the evening for six consecutive days.
  Interventions: Device: Mandala
- control group (No Intervention): The control group will receive the usual care.

INTERVENTIONS:
Device: Mandala — Experimental group will paint mandala for 30 minutes/day in the evenings for six consecutive days. Six pre-selected mandalas were planned to be printed separately on A4 paper. Each patient will be given a new mandala each day. Additionally, At the beginning of the study, the experimental group will be given six colors (yellow, blue, green, red, purple, brown).
  Other Names: Mandala Painting
  Arms: intervention group

SUMMARY:
This study was planned as a randomized controlled trial to determine the effect of mandala painting on the anxiety of coronary heart patients.

DETAILED DESCRIPTION:
Patients in the control group will receive routine care.Patiens in the experimental group will receive routine care and mandala painting. Experimental group will paint mandala for 30 minutes/day in the evenings for six consecutive days. In order not to interrupt the duties of the nurse and doctor in the clinic, it was planned for the experimental group to paint mandalas in the evening. Six pre-selected mandalas were planned to be printed separately on A4 paper. Each patient will be given a new mandala each day. At the beginning of the study, six colors will be given to the experimental group (yellow, blue, green, red, purple, brown). It was planned to do it for 6 days, as it was found that painting mandala for more than a week in the studies could reduce the patient's attention. In addition, based on the average hospitalization days of the patients, reaching patients for more than a week will be a problem.

ELIGIBILITY:
Inclusion Criteria:

* Having agreed to participate in the research/approved the informed consent form
* No visual or hearing impairment
* Hospitalization due to Coronary Heart Disease (patients hospitalized with the diagnosis of acute coronary syndromes such as stable angina, unstable angina, myocardial infarction, percutaneous coronary intervention and stent implantation),
* Being over 18 years old,
* Being at least literate
* The absence of any problem that would prevent him/her from painting mandala (no problem in his arm or hand that would prevent his movement (such as paralysis, or the presence of a catheter on the hand), no serious illness)
* Must not have a diagnosis of mental illness/anxiety disorder

Exclusion Criteria:

* Control group patients who coincided with the same room as the intervention group, by randomization.
* Patients who want to quit the study voluntarily during the study
* Patients whose general condition deteriorates (such as altered hemodynamics or consciousness)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-09 (Actual); Primary Completion 2023-08-09 (Actual); Study Completion 2023-09-23 (Actual)

PRIMARY OUTCOMES:
The Hospital Anxiety and Depression Scale | six days
  The scale consists of 14 items including 7 anxiety and 7 depression questions. Responses are in the form of a four-point likert. Each item is scored between 0 and 3, and the cut-off points of the scale were found to be 10 for the anxiety subscale and 7 for the depression subscale. Individuals who score above these scores are considered at risk. The scoring score of each item in the scale is different, and the 1st, 3rd, 5th, 6th, 8th, 10th, 11th and 13th items show that the severity is gradually decreasing and its scoring is 3, 2, 1, 0. The 2nd, 4th, 7th, 9th, 12th and 14th items of the scale are scored as 0, 1, 2, 3. Items 1, 3, 5, 7, 9, 11, and 13 for the anxiety subscale, and items 2, 4, 6, 8, 10, 12, and 14 for the depression subscale. The scores of the items are summed. The lowest zero and the highest 21 points can be obtained from both sub-dimensions of the scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Çamcı, PhD, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No